CLINICAL TRIAL: NCT02873403
Title: A 3D Printed Knee Brace to Improve Symptoms, Biomechanics and Daily Life Among Medial Knee Osteoarthritis Patients
Brief Title: Novel 3D Printed Knee Brace for Medial Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peacocks Medical Group (Industry)
Collaborators: Glasgow Caledonian University (Other); Universität Münster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AMKNEEBRACE01
Record Dates: First submitted 2016-07-27; First posted 2016-08-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KNEEMO knee brace & Popular knee brace (Experimental): Patients having medial knee osteoarthritis
  Interventions: Device: KNEEMO knee brace; Device: Popular knee brace
- Popular knee brace &KNEEMO knee brace (Experimental): Patients having medial knee osteoarthritis
  Interventions: Device: KNEEMO knee brace; Device: Popular knee brace

INTERVENTIONS:
Device: KNEEMO knee brace — Bespoke knee brace made by additive manufacturing
Device: Popular knee brace — Customized knee brace used in the management of medial knee ostearthritis

SUMMARY:
Around 250 millions of people in the world (3.8%) have knee osteoarthritis (KOA). Due to aging and increasing obesity, the prevalence of KOA is expected to increase in the developed country in the next 20 years. KOA decreases quality of life of patients through chronic pain, joint stiffness, and reduced social activity, which influence emotional wellness as well. KOA has also impact on the biomechanics of the lower limbs, leading or amplifying the tibiofemoral misalignment and an increase of the medial knee joint loading. Increase of the medial knee joint loading may lead patients into a vicious circle by increasing knee pain, decreasing activities, increasing weight and disease progression. Knee brace is a non-pharmacological treatment recommended for KOA. It aims to reduce misalignment of the limb. However, the main issue is the poor compliance because of lack of effectiveness, more drawbacks than benefits, discomfort, bad fitting, migration of the brace, bulkiness, aesthetic, skin irritation, blisters and too much pressure on the knee. By its freedom in design, 3D printing may resolve most of these complaints.

This study aims to compare clinical and biomechanical effectiveness, comfort and patients complaints of a knee brace made by 3D printing to a conventional knee brace.

The institute for Applied Health Research of Glasgow Caledonian University (GCU) will lead the experimental trial. They will recruit men or women (40 to 70 years old) suffering from medial KOA in Glasgow area. Participants will be in study for 10 weeks. During this period, they will wear 2 different knee braces for two weeks each with a 1-week period without knee brace between. Participants will have five visits to GCU: once for leg measurement to make knee braces and four times to fill questionnaires and perform gait analysis. Besides, they will wear activity monitor for 3 non-consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 40 and 70 years old having radiological and symptomatic medial KOA (Kellgren-Lawrence grade II, III or IV) according to the American College of Rheumatology's clinical and radiological criteria [83]
* Average knee pain > 4/10 (VAS score assessed three times in two weeks before being included)
* Not currently wearing knee brace
* Varus knee alignment equal or superior to 2°
* No or light pain from the hips, ankles, feet or lumbar spine
* Moderately physically active
* Able to understand written and spoken English.

Exclusion Criteria:

* Mild KOA (Kellgren-Lawrence grade I)
* Lateral or patellar KOA
* Chronic diseases or conditions (e.g., diabetes, osteoporosis, heart disease, hypertension, neurological disorders)
* Stroke history
* Inflammatory arthritis (gout, RA, psoriatic arthritis, …)
* Musculoskeletal disorders that could influence their ability to stand and walk
* Morbid obesity (BMI > 35)
* Intra-articular corticosteroid/hyaluronan injection in the affected knee in the past 3 months
* Unstable medication schedule and medication that causes dizziness
* Severe recent modification of diet
* Prosthetic implants in the hip, knee or ankle joint
* Poor skin condition
* Unable to walk, walk up and down stairs or any condition contraindicating the demands of the gait analysis.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in knee pain during gait and stairs ambulation | Baseline and at 2 weeks
  Measured with 10-cm visual analog scale
Change in knee adduction moment during gait and stairs ambulation | Baseline and at 2 weeks
  Knee adduction moment (KAM) will be calculated from motion capture and force plate data. KAM characterizes knee loading, especially peaks and angular impulse (area under the KAM curve) to have information about maximum and total knee loading, respectively.

SECONDARY OUTCOMES:
Change in knee brace comfort | Baseline and at 2 weeks
  Measured with 10-cm visual analog scale
Change in stability feelings | Baseline and at 2 weeks
  Measured with 10-cm visual analog scale
Change in Symptoms | Baseline and at 2 weeks
  KOOS questionnaires subscales
Change in quality of life | Baseline and at 2 weeks
  MOS SF-36 questionnaires subscales
Change in physical activities: Daily distance estimate | Second week of intervention
  Measured (in km) during one week with an activity monitor.
Change in physical activities: Daily duration of sitting/standing/stair climbing | Second week of intervention
  Measured in seconds during one week with an activity monitor.
Change in physical activities: Daily number of sitting/standing/stair climbing | Second week of intervention
  Measured during one week with an activity monitor.
Change in physical activities: Weekly number of activities with moderate and high intensity | Second week of intervention
  Measured during one week with an activity monitor.
Change in physical activities: Weekly duration of activities with moderate and high intensity | Second week of intervention
  Measured in minutes during one week with an activity monitor.
Change in knee flexion moment during gait and stairs ambulation | Baseline and at 2 weeks
  Maximum knee flexion moment will be calculated from gait analysis data.
Change in duration of phases of gait and stairs ambulation | Baseline and at 2 weeks
  Measured in percentage of gait cycle from gait analysis data.
Change in step length of gait | Baseline and at 2 weeks
  Measured in meters from gait analysis data
Change in knee flexion/extension range of motion during gait and stairs ambulation | Baseline and at 2 weeks
  Measured during the gait cycle based on gait analysis data
Change in knee adduction/abduction range of motion during gait and stairs ambulation | Baseline and at 2 weeks
  Measured during the gait cycle based on gait analysis data

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Dessery, PhD, Principal Investigator — Peacocks Medical Group
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom